CLINICAL TRIAL: NCT05345067
Title: The Effect of Laughter Yoga on the Anxiety and Stress Levels of Women in the Postpartum Period: A Randomized Controlled Trial
Brief Title: The Effect of Laughter Yoga on the Anxiety and Stress Levels of Women in the Postpartum Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Aslı SİS ÇELİK, Associate Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: aslı25
Record Dates: First submitted 2022-04-19; First posted 2022-04-25 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Laughter Yoga
Keywords: Laughter Yoga; Postpartum Period; Anxiety; Stress; Nurse
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: The women in the experimental and control groups did not know which group they were in. Data were collected online due to the pandemic. Therefore, the researchers and the people who would conduct the analyzes did not know the women in the experimental and control groups. The women used a nickname to fill in the questions on the measurement tools.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental: Laughter yoga session parts-1 (Experimental): Deep breathing exercises (5 minutes)
  Interventions: Behavioral: Experimental: Laughter yoga session parts-1
- Experimental: Laughter yoga session parts-2 (Experimental): Warm-up exercises (10 minutes)
  Interventions: Behavioral: Experimental: Laughter yoga session parts-2
- Experimental: Laughter yoga session parts-3 (Experimental): Childish games (10 minutes)
  Interventions: Behavioral: Experimental: Laughter yoga session parts-3
- Experimental: Laughter yoga session parts-4 (Experimental): Laughter exercises (15 minutes)
  Interventions: Behavioral: Experimental: Laughter yoga session parts-4

INTERVENTIONS:
Behavioral: Experimental: Laughter yoga session parts-1 — Section 1: Deep breathing exercises: A deep breath is taken as far as possible by raising the arms up to the sky. Breathing is held for 4-5 seconds after deep inspiration. Breathing is performed rhythmically and slowly, while the arms are placed in a normal position. After deep inspiration, one can exhale either by forming the lips in the whistling position or by laughing. In each deep breathing exercise technique, the expiration time of the exhalation process should be longer than the inspiration time.
  Arms: Experimental: Laughter yoga session parts-1
Behavioral: Experimental: Laughter yoga session parts-2 — Section 2: Warm-up exercises (10 minutes): Hands are clapped by holding parallel to each other. The fingertips and the palms touch each other, stimulating the acupuncture points on both hands, and the individual's energy level rises. In order to further raise the energy level and synchronize the movements of the group, a rhythm is added in the form of 1-2, 1-2-3. After several rhythmic hand-clapping movements, one more movement is added. Hands are clapped by swinging left and right. Then, an audible rhythm in the form of ho, ho, ha-ha-ha is also added to the hand-clapping movement. People in the group look at each other, and smile.
  Arms: Experimental: Laughter yoga session parts-2
Behavioral: Experimental: Laughter yoga session parts-3 — Section 3: Childish games (10 minutes): Childish games are used that will help to laugh for no reason, just like a child. Imagining these games and plays, the arms are raised upwards in the form of a "Y" with palms facing the sky, motivating the group by saying "very good (clap), very good (clap), yes". The leader of laughter yoga speaks out "very good (clap), very good (clap), hey (arms to the right and left)" to keep the group's energy high and generate enthusiasm in the deep breathing exercises and laughter exercises sections. According to the energy and desire of the group, this section is completed after about 10 minutes.
  Arms: Experimental: Laughter yoga session parts-3
Behavioral: Experimental: Laughter yoga session parts-4 — Section 4: Laughter exercises (15 minutes): This section contains a variety of laughter exercises that will laugh, such as greetings, laughter cream, exploding balloon laughter, preparing and drinking strawberry milk, bonuses, hot soup, lion, aloha, bird, appreciation, elevator, and cream pie. A laugh is raised by doing only laughter exercises for no reason at all. At the end of this section, relaxation is achieved for about three minutes using deep breathing exercises. The group is given verbal guidance "Put your hand on your heart, feel your heartbeat, let's exhale with a smile, make a wish or pray, smile as if we had achieved our wish," and the laughter yoga session is terminated.
  Arms: Experimental: Laughter yoga session parts-4

SUMMARY:
This research is a randomized controlled study to evaluate the effect of Laughter yoga on the anxiety and stress levels of postpartum women. Randomization was provided in the sample included in the study, and it was divided into experimental and control groups. At the beginning of the study, the Postpartum anxiety scale and the perceived stress scale were applied to women in both groups to determine their anxiety and stress levels. Afterwards, 8 sessions of laughter yoga were applied to the experimental group for 4 weeks. No application was made to the control group. After 4 weeks, the Postpartum anxiety scale and the perceived stress scale were administered to the women in both groups to re-determine their anxiety and stress levels.

DETAILED DESCRIPTION:
This research is a randomized controlled study to evaluate the effect of Laughter yoga on the anxiety and stress levels of postpartum women. At the beginning of the study, necessary ethics committee permission and institutional permissions were obtained. Both of the researchers have a certificate of leadership in laughter yoga. As a result of the power analysis, it was determined that 128 women should be included in the study. Considering that there may be losses, it was decided to include 160 women in the study. By providing randomization, 160 women who met the sampling criteria and volunteered to participate in the study were divided into two groups as 80 experimental and 80 control. At the beginning of the study, the Postpartum anxiety scale and the perceived stress scale were applied to women in both groups to determine their anxiety and stress levels. Afterwards, 8 sessions of laughter yoga were applied to the experimental group for 4 weeks, two sessions a week. No application was made to the control group. After 4 weeks, the Postpartum anxiety scale and the perceived stress scale were administered to the women in both groups to re-determine their anxiety and stress levels. In the study, 7 women from the experimental group and 9 women from the control group were excluded for various reasons. The study was conducted with 73 experimental and 71 control groups. The process of making analyzes and writing the final report continues. This study is financially supported by Atatürk University Scientific Research Coordination Unit. In addition, this study is carried out as a master's thesis accepted by Atatürk University Health Sciences Institute.

ELIGIBILITY:
Inclusion Criteria:

* be between the ages of 19-45
* Giving birth by vaginal / Caesarean section
* 1 month after birth
* Having a healthy baby
* Not experiencing any complications during birth and postpartum
* At least primary school graduate
* Not having a diagnosed psychiatric disease

Exclusion Criteria:

* Having a medical condition (hypertension, wound complication, etc.)
* Not regularly attending laughter yoga sessions (for the experimental group)
* Applying another alternative method to reduce anxiety and stress in the postpartum period

Ages: 19 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Questionnaire Form | up to 2 weeks
  Prepared by the researcher; There are introductory information such as age, education level, family type and 24 questions about the postpartum period. This form determines the introductory characteristics of the participants. therefore no points are taken.
Postpartum Specific Anxiety Scale | up to 2 weeks
  This scale was developed by Fallon et al. to evaluate postpartum anxiety symptoms. The Turkish adaptation of the scale was made by Duran in 2019. Since it was determined that some items could be in different groups in the adaptation to Turkish, it was decided to be one-dimensional and some items not to be in the Turkish version. The Turkish form of the scale was evaluated as one-dimensional and 47 items. It can be said that those who score 73 and below on the scale have low postpartum anxiety levels, those who score between 74 and 100 have a medium level, and those who score 101 and above have a high level of anxiety.
Perceived Stress Scale | up to 2 weeks
  It was developed by Cohen, Kamarck & Mermelste in 1983 to measure the perceived stress of a person in any situation, and was adapted into Turkish by Eskin et al. It contains 14 items in total. Participants evaluated the items on a 5-point Likert-type scale ranging from "Never (0)" to "Very often (4)". 7 items containing positive statements are scored in reverse. Scoring ranges from 0 to 56, while a high score indicates that the person is highly stressed.

SECONDARY OUTCOMES:
Postpartum Specific Anxiety Scale | up to 3 weeks
  This scale was developed by Fallon et al. to evaluate postpartum anxiety symptoms. The Turkish adaptation of the scale was made by Duran in 2019. Since it was determined that some items could be in different groups in the adaptation to Turkish, it was decided to be one-dimensional and some items not to be in the Turkish version. The Turkish form of the scale was evaluated as one-dimensional and 47 items. It can be said that those who score 73 and below on the scale have low postpartum anxiety levels, those who score between 74 and 100 have a medium level, and those who score 101 and above have a high level of anxiety.
Perceived Stress Scale | up to 3 weeks
  It was developed by Cohen, Kamarck & Mermelste in 1983 to measure the perceived stress of a person in any situation, and was adapted into Turkish by Eskin et. It contains 14 items in total. Self-efficacy and perception of stress It consists of two sub-dimensions. Participants evaluated the items on a 5-point Likert-type scale ranging from "Never (0)" to "Very often (4)". 7 items containing positive statements are scored in reverse. Scoring ranges from 0 to 56, while a high score indicates that the person is highly stressed.

CONTACTS AND LOCATIONS:
Overall Officials: Aslı SİS ÇELİK, Study Director — Ataturk University
Locations (1):
- Atatürk University, Erzurum, Yakutiye, Turkey (Türkiye)